CLINICAL TRIAL: NCT04749212
Title: Incidence and Clinical Relevance of Perioperative Elevation of Troponin I and N- Terminal Pro-Brain Natriuretic Peptide in Patients Undergoing Lung Resection
Brief Title: Perioperative Troponin I and NT Pro-BNP in Lung Resection
Status: Completed | Type: Observational
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 621/2020
Record Dates: First submitted 2021-01-18; First posted 2021-02-11 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Cardiac Ischemia; Thoracic Cancer; Complication,Postoperative
MeSH Terms: conditions — Coronary Artery Disease; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: serum high-sensitivity Troponin I (TnI) and NT-Pro-Brain Natriuretic Peptide (NT-proBNP) — Both biomarkers will be determined in each patient preoperatively and at postoperative day 1 and day 2.Measurements will not necessarily be taken independently of other measurements, meaning that the addition of the biomarker could be included in routine pre or postoperative day-1 and day 2 blood tests.

SUMMARY:
After lung resection, troponin elevation may be regulated by mechanisms other than myocardial ischemia. Perioperative natriuretic peptides measurement may help identify changes in ventricular function during thoracic surgery. Integrating both cardiac biomarkers may improve the predictive value for cardiovascular complications after lung resection.

DETAILED DESCRIPTION:
Objectives: To evaluate the incidence and magnitude of perioperative N-terminal pro brain natriuretic peptide (NT-proBNP) and high-sensitivity troponin I (Tn I) elevation in patients undergoing pulmonary resection and its predictive value for cardiovascular complications. Methodology: Prospective, multicenter, observational cohort study in patients >45 years undergoing elective thoracic surgery for lung resection. Cardiac biomarkers Tn I and NT-proBNP will be measured preoperatively and at postoperative days 1 and 2. Risk score for major cardiovascular postoperative complications will be calculated depending of both biomarkers perioperative changes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥45 years old
* Patients undergoing elective surgery for lung resection

Exclusion Criteria:

* Patients undergoing urgent, emergent, or nonthoracic surgery
* Patients or family did not consent to participate
* Presence of symptoms related with infection or sepsis
* Patients with a documented history of severe heart failure and/or ejection fraction lower than 30%

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adulty patients undergoing elective thoracic and lung resection surgery: neumonectomy, lobectomy, bilobectomy or segmentectomy
Sampling Method: Non-Probability Sample
Enrollment: 475 (Actual)
Dates: Start 2021-05-19 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
NT-proBNP perioperative changes | Change from baseline NT-proBNP at two-days after surgery
  Perioperative change in NT-Pro-Brain Natriuretic Peptide (NT-proBNP) levels in patients undergoing pulmonary resection. Cutt-of values will be NT-proBNP ≥ 300 pg/ml pg/ml
TnI perioperative changes | Change from baseline TnI at two-days after surgery
  Perioperative changes in high-sensitivity troponin I (TnI) levels in patients undergoing pulmonary resection. Cutt-of values will be TnI ≥45 ng/L
Major cardiovascular complications | 30-days after surgery
  Postoperative non-fatal cardiac arrest, acute myocardial infarction, angina, congestive heart failure, new clinically relevant cardiac arrhythmia, cardiovascular death

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari Vall d'Hebron, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alonso M, Popova E, Martin-Grande A, Perez-Velez J, Trujillo JC, Gajate L, de Miguel M, Gonzalez-Tallada A, Martinez-Tellez E, Cladellas-Gutierrez E, Planas G, de Pablo A, Parise D, Candela-Toha A, de Nadal M. Study protocol for an observational cohort evaluating incidence and clinical relevance of perioperative elevation of high-sensitivity troponin I and N-terminal pro-brain natriuretic peptide in patients undergoing lung resection. BMJ Open. 2022 Dec 8;12(12):e063778. doi: 10.1136/bmjopen-2022-063778. PMID 36600389